CLINICAL TRIAL: NCT06677710
Title: A Phase 1B Study of IDP-023 g-NK Cells Plus Ocrelizumab in Patients With Refractory Primary and Secondary Progressive Multiple Sclerosis
Brief Title: IDP-023 g-NK Cells Plus Ocrelizumab in Patients With Progressive Multiple Sclerosis
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Indapta Therapeutics, INC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDP023-2-101
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Primary Progressive Multiple Sclerosis (PPMS); Secondary Progressive Multiple Sclerosis (SPMS); Non-Active Secondary Progressive Multiple Sclerosis; Non-Active SPMS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Autoimmune Diseases; Demyelinating Diseases; Immune System Diseases; Demyelinating Autoimmune Diseases, Central Nervous System (CNS)
Keywords: Progressive Multiple Sclerosis; Refractory Progressive Multiple Sclerosis; IDP-023; autoimmune disease; Cellular Therapy; MS; Natural Killer Cells
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Autoimmune Diseases; Demyelinating Diseases; Immune System Diseases; Demyelinating Autoimmune Diseases, CNS | interventions — ocrelizumab; Interleukin-2; aldesleukin; Cyclophosphamide; fludarabine; Mesna

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose and dose-expansion study of IDP-023 in combination with interleukin-2 (IL-2) and ocrelizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (dose escalation): IDP-023 in combination with IL-2 and ocrelizumab (Experimental): MS patients treated with multiple doses of IDP-023 in combination with IL-2 and ocrelizumab
  Interventions: Drug: IDP-023; Drug: Ocrelizumab; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Part 2 (dose expansion): IDP-023 in combination with IL-2 and ocrelizumab (Experimental): MS patients treated with the recommended dose of IDP-023 in combination with IL-2 and ocrelizumab
  Interventions: Drug: IDP-023; Drug: Ocrelizumab; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna

INTERVENTIONS:
Drug: IDP-023 — NK cell therapy
Drug: Ocrelizumab — Anti-CD20 antibody therapy
  Other Names: Ocrevus
Drug: Interleukin-2 — Immune cytokine
  Other Names: Proleukin
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy
Drug: Mesna — Chemoprotectant

SUMMARY:
This is an open label, Phase 1b, multiple ascending dose, and dose-expansion study of IDP-023 administered in combination with interleukin-2 (IL-2) and ocrelizumab to evaluate the safety, tolerability, and biologic activity on autoreactive immune cells in patients with refractory progressive multiple sclerosis.

DETAILED DESCRIPTION:
IDP-023 is an off-the-shelf product made from allogeneic g-natural killer (NK) cells, which are a natural subset of NK cells that develop over the course of an immune response in people who have been exposed to the human cytomegalovirus (HCMV). These cells may be particularly effective at targeting and killing the cells that cause the immune system to attack the nervous system in multiple sclerosis (MS). By killing these harmful cells, g-NK cells may help to slow down or potentially stop the progression of MS. When combined with other approved treatments like ocrelizumab, g-NK cells might offer even greater beneﬁt for people with MS.

This is an open label, Phase 1b, multiple ascending dose, and dose-expansion study of IDP- 023 administered in combination with IL-2 and ocrelizumab to evaluate the safety, tolerability, and biologic activity on autoreactive immune cells in patients with primary progressive multiple sclerosis (PPMS) or non-active secondary progressive multiple sclerosis (SPMS).

The study is divided into Part 1, a dose escalation phase, and Part 2, an expansion phase.

Part 1 (Escalation Period): The primary objectives of Part 1 are to deﬁne the safety of different dose levels of IDP-023 in combination with IL-2 and ocrelizumab and to deﬁne the recommended cell dose that will be used for Part 2 (recommended Part 2 dose; RP2D).

Part 2 (Expansion Period): The objective of the Part 2 expansion phase is to assess the biologic activity of IDP-023 in combination with IL-2 and ocrelizumab on autoreactive immune cells in PPMS.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of primary or non-active secondary progressive MS (SPMS) based on the 2017 revisions of the McDonald criteria.
* Dosed with ocrelizumab within the prior 6 months.
* Expanded Disability Status Scale (EDSS) at screening from 3.0 to 6.5 points.
* Score of ≥2.0 on the Functional Systems (FS) scale for the pyramidal system that is due to lower extremity findings.
* Disease duration from the onset of MS symptoms:

  * Less than 15 years in patients with an EDSS at screening >5.0.
  * Less than 10 years in patients with an EDSS at screening ≤5.0.

Key Exclusion Criteria:

* Relapsing remitting MS at screening or active SPMS at screening.
* Inability to complete an MRI.
* Contraindication for gadolinium.
* Known presence of other neurological disorders, including but not limited to the following:

  * History or known presence of CNS or spinal cord tumor (e.g., meningioma, glioma).
  * History or known presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, Human T-lymphotropic virus 1 [HTLV-1], herpes zoster myelopathy).
  * History or known presence of systemic autoimmune disorders potentially causing progressive neurologic disease (e.g., lupus, antiphospholipid antibody syndrome, Sjögren's syndrome, Behçet's disease).
* Impaired cardiac function or history of clinical significant cardiac disease.
* Human immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs - (Part 1) | 1 year
  Escalation Period
Incidence of dose-limiting toxicities (DLTs) of IDP-023 in combination with IL-2 and Ocrelizumab (Part 1) | up to 21 days
  Escalation Period
Change in cellular response of autoreactive immune cells to antigen (Part 2) | 2 years
  Expansion Period

SECONDARY OUTCOMES:
Change in cellular response of autoreactive immune cells to antigen (Part 1) | 2 year
  Escalation Period
Incidence of AEs and SAEs - (Part 2) | 2 years
  Expansion Period
PK (PK; maximum drug concentration) of IDP-023 - (Part 1/2) | 2 years
  Escalation and Expansion periods
PK (area under the concentration-time curve) of IDP-023 - (Part 1/2) | 2 years
  Escalation and Expansion periods
PK (concentration reached by the drug immediately before the next dose is administered) of IDP-023 - (Part 1/2) | 2 years
  Escalation and Expansion periods
Time to onset of sustained disability progression over the treatment period, deﬁned as an increase in Expanded Disability Status Scale (EDSS) - (Part 1/2) | 2 years
  Escalation and Expansion periods
Biologic activity of IDP-023 in the CSF over the treatment period - (Part 1/2) over the treatment period, defined as an increase in EDSS - (Part 1/2) | 2 years
  Escalation and Expansion periods

CONTACTS AND LOCATIONS:
Overall Officials: Indapta Therapeutics, Inc., Study Director — Indapta Therapeutics, INC.
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - AdventHealth Orlando - Adventist Health System/Sunbelt, Inc., Orlando, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No